CLINICAL TRIAL: NCT04869553
Title: Analgesic Efficacy of Hypnosis and Virtual Reality in Repetitive Pain Care : a Controlled, Randomised, Cross-over, Open-label, Multi-centre Study
Brief Title: Analgesic Efficacy of Hypnosis and Virtual Reality in Repetitive Pain Care
Acronym: PADIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: RC-P00102
Record Dates: First submitted 2021-04-28; First posted 2021-05-03 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Pain
Keywords: Pain management; Hypnosis; Virtual Reality; Distractibility methods
MeSH Terms: conditions — Pain; Agnosia | interventions — Analgesia

STUDY DESIGN:
Intervention Model Description: Controlled, randomised, open-label, cross-over, 3-sequence study (uniform design across time and sequence: ABC/BCA/CAB).
  * Treatment A: Usual pain management of each ward
  * Treatment B: Usual pain management on each ward and analgesic hypnotherapy during care
  * Treatment C: Usual pain management of each ward and virtual reality session using a suitable headset.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- ABC's arm (Experimental): The 3 pain managements are in the ABC's order.
  Interventions: Other: Management pain with distraction methods ABC
- BCA's arm (Experimental): The 3 pain managements are in the BCA's order.
  Interventions: Other: Management pain with distraction methods BCA
- CAB's arm (Experimental): The 3 pain managements are in the CAB's order.
  Interventions: Other: Management pain with distraction methods CAB

INTERVENTIONS:
Other: Management pain with distraction methods ABC — Every patient will receive :
  * The usual pain management of their ward (Treatment A),
  * The usual pain management of their ward with a hypnosis session (Treatment B)
  * The usual pain management of their ward with a virtual reality session (Treatment C)
  Arms: ABC's arm
Other: Management pain with distraction methods BCA — Every patient will receive :
  * The usual pain management of their ward with a hypnosis session (Treatment B)
  * The usual pain management of their ward with a virtual reality session (Treatment C)
  * The usual pain management of their ward (Treatment A)
  Arms: BCA's arm
Other: Management pain with distraction methods CAB — Every patient will receive :
  * The usual pain management of their ward with a virtual reality session (Treatment C)
  * The usual pain management of their ward (Treatment A)
  * The usual pain management of their ward with a hypnosis session (Treatment B)
  Arms: CAB's arm

SUMMARY:
The originality of this study is the comparison of different distractibility techniques (hypnosis and virtual reality) in the very heterogenous contexts of pain management. This study will consider all types of care situations. The study's cross-over design will take into account this heterogenous context. The results will be representative of real-life situations where care for pain involves a wide range of contexts.

DETAILED DESCRIPTION:
Pain is defined as an unpleasant sensorial and emotional experience related to a potential or existing tissue injury (psychological (affective) and physical dimension of pain). Since it can occur at any stage of care, pain concerns all healthcare teams working in acute care units or follow-up care centers.

At the present time, pain management is mainly based on the use of analgesic agents that calm or suppress pain. Different types of analgesic agents are available in the therapeutic armamentarium (non-opioid analgesics and opioid analgesics as morphine).

In this context where pain management is a priority and where the use of morphine is constantly on the rise exposing patients to significant risk (adverse effects, addictions, respiratory events….), the use of distractibility techniques as hypnosis and virtual reality could be an attractive alternative.

* Hypnosis designates both a therapeutic technique and a modified state of consciousness also called trance (a state where the person is between a state of wakefulness and sleep).
* Virtual reality designates a three-dimensional computer-controlled environment allowing immersion, interaction and multisensorial input.

Thus, the originality of this study is the comparison of different distractibility techniques in the very heterogenous contexts of pain management. This study will consider all types of care situations. The study's cross-over design will take into account this heterogenous context. The results will be representative of real-life situations where care for pain involves a wide range of contexts.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing care interventions of a given type (e.g. wound dressings/mobilization/…) recognized as painful (pain VAS >3 despite the usual analgesic protocol)
* Repetition of the same type of intervention at least three times within a month of interval after inclusion
* Patient age ≥15 years
* Informed consent from patient or legal guardian
* Beneficiary of the French healthcare fund

Exclusion Criteria:

* MEOPA's administration during painful treatment as part of the study
* Cognitive or psychiatric disorders preventing the patient from communicating with caregivers or understanding their instructions
* Any other concomitant nervous system, cardiac, or pulmonary disease that might affect the autonomous nervous system: (myocardial infarction, myocardial disorder (e.g. dilated or hypertrophic cardiomyopathy), class 3 or 4 heart failure, cardia dysrhythmia, including atrial fibrillation, conduction disorder, mechanical ventilation)
* Non-sinusal rhythm, extrasystoles, altered ECG signals related to heart disease
* Mandatory drug therapy that might affect the autonomous nervous system and NRV such as beta-blockers, muscarinic receptor blockers (mainly atropine, scopolamine), vasopressin agents
* Contraindication for use of the virtual reality headset and/or hypnosis. Neurological disorder incompatible with use of the virtual reality headset and/or hypnosis (balance disorders/seizures…)
* Contraindication for using surface electrodes preventing collection of the main endpoint data
* Any disorder or disability preventing execution of the virtual reality or hypnosis techniques (deafness/blindness)
* Judicial protection status

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-01-07 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-05-24 (Actual)

PRIMARY OUTCOMES:
Analgesia Nociception Index (ANI) during painful care interventions | one month
  This index is derived from heart rate variability and reflects the relative parasympathetic tone. An ANI value close to 100 corresponds to a prominent parasympathetic tone (low stress level, analgesia) and a value close to 0 corresponds to a prominent sympathetic tone (high stress level, nociception).

SECONDARY OUTCOMES:
ANI's average score (Analgesia Nociception Index) 5 minutes after the care and the distractibility methods | one month
  A comparison between the ANI's score before and after the care and the distractibility methods. The average of the scores will be retained.
Visual Analog Scale (VAS) | one month
  The pain's level will be evaluated by the Visual Analog Scale (VAS). This scale measure the pain's intensity from 0 to 10.
Morphine equivalent | one month
  The opioid analgesics administered during the care will be converted into morphine equivalent by means of the opioid equi-analgesia table. The collection of analgesics will include all analgesics "in action" on the day of care.
Proportion of patients tolerance to distractibility techniques | one month
  All events leading to a discontinuation of the distractibility technique will be recorded: side effects /cybersickness (nausea, vertigo evaluated using the Speech, Spatial and Qualities (SSQ) of Hearing Scale prolonged procedure, dissociative disorders …), patient refusal, care-related elements preventing the use of the distractibility technique or leading to premature discontinuation of its use.
Correlation between patient age and tolerance | one month
  The impact of age on abandon (irrespective of the reason) will be noted to search for a link between age and tolerance.
Correlation between patient age and treatment efficacy | one months
  The impact of age on treatment effect on ANI score during the care procedure will be noted to search for a link between age and treatment efficacy.
Correlation between caregiver training level and hypnosis efficacy | one month
  Hypnosis training level will be determined by the duration of training (hours) and the professional level (1/2/3). Caregiver category (nurse/psychologist/rehabilitation specialist…) and the number of hypno-therapy sessions delivered during the six months preceding the study will also be considered.
Percentage of satisfaction concerning the distractibility techniques. | one month
  A questionnaire will evaluate patient perceptions concerning the distractibility techniques.
IPQ (Igroup Presence Questionnaire) scale | one month
  The IPQ is a 14-item self-administered questionnaire. This scale is used to measure the patient's feelings about spatial presence, the implication and sense of the reality perceived in the virtual reality.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Noëlle BARTHOLOMEI, PharmD, Study Director — Hôpital Léon Bérard
Locations (5):
- France (5):
  - Hôpital Léon Bérard, Hyères
  - USSAP - Centre Bouffard Vercelli, Perpignan
  - Centre Mutualiste de Kerpape, Ploemeur
  - Pôle MPR Saint Hélier, Rennes
  - Fondation ILDYS - Site de Perharidy, Roscoff

IPD SHARING:
Plan to Share IPD: No